CLINICAL TRIAL: NCT04735406
Title: The MS-LINK™ Outcomes Study: A Comprehensive Prospective Longitudinal Assessment of Patient and Clinical Reported Outcomes in Multiple Sclerosis Patients Across North America
Brief Title: The MS-LINK™ Outcomes Study
Status: Completed | Type: Observational
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS200077_0021
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: Expanded Disability Status Scale; Multiple Sclerosis; Patient Reported Outcomes Measurement Information System
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Sclerosis (MS): Data from the participants with diagnosed MS treated and untreated will be part of this study. Medical records of participants will be used to collect demographics and data pertaining to Multiple Sclerosis (MS) management.

SUMMARY:
The Multiple Sclerosis (MS) Leadership and Innovation Network (MS-LINK™) is comprised of networks working cooperatively to advance Multiple Sclerosis (MS) science and improve MS participant outcomes. In this study participants will be followed from the time of consent through the lifetime of the study (currently 3 years), unless the participant chooses to withdraw from the study. Collection of participant's medical history, including MS and treatment history, will be automated through extraction from the participant's electronic medical record (EMR) and other health information systems (for example, radiology). Participants will complete patient-reported outcomes (PROs) and other health-related information digitally. Participating participants will have access to their own data in an ongoing manner via a web-based Participant Portal.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide written informed consent
* Participants willing to be contacted while participating in the study for recruitment into sub-studies that may be relevant to them
* Participants willing and able to complete PROs on a monthly basis and document events of interest as they occur
* Participants willing to participate in additional follow up at the site for at least three years

Exclusion Criteria:

* Unable to complete questionnaires in English
* Unable to consistently access the Internet
* Participants participating in interventional clinical drug trials at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from United states and Canada with Multiple sclerosis (MS) will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2182 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Patient-determined Disease Steps (PDDS) Scale Score | Baseline up to 3 years
Patient Reported Outcomes Measurement Information System (PROMIS) Multiple Sclerosis (MS) Fatigue Score | Baseline up to 3 years
Patient Reported Outcomes Measurement Information System (PROMIS) Multiple Sclerosis (MS) Physical Function Score | Baseline up to 3 years
Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Score | Baseline up to 3 years
Patient Reported Outcomes Measurement Information System (PROMIS) MS Cognitive Function Score | Baseline up to 3 years
Patient Health Questionnaire 9-Item (PHQ9) Score | Baseline up to 3 years
Wasson Health Confidence Scale Score | Baseline up to 3 years
Health-related Quality of Life Assessed by Centers for Disease Control and Prevention Health-Related Quality of Life Measure (CDC HRQoL-14) | Baseline up to 3 years
Work Productivity and Activity Impairment Questionnaire-Multiple Sclerosis (WPAI-MS) Score | Baseline up to 3 years
Number of Participants with Reasons for Discontinued Disease-Modifying Therapies (DMT) | Baseline up to 3 years
Number of Participants with Current Use of Disease-Modifying Therapies (DMT) | Baseline up to 3 years
Duration of Disease-Modifying Therapies (DMT) use | Baseline up to 3 years
Number of Participants With Adherence to Treatment as Assessed by Multiple Sclerosis Treatment Adherence Questionnaire (MS-TAQ) | Baseline up to 3 years
Occurrence of Relapses | Baseline up to 3 years
Occurrence of Multiple Sclerosis (MS) Symptoms | Baseline up to 3 years
Number of Utilization of Healthcare Resources by Participants | Baseline up to 3 years
Well-being of Participant Assessed by Physical Activity Diary | Baseline up to 3 years
  Participants can opt-in to use the Patient Portal to track their well-being in up to 9 domains like Sleep, Mood, Pain, Exercise, Mobility, Wellness, Energy, Bladder Function, Leisure activities.
Number of Participants with Response to Health Priorities and Goals | Baseline up to 3 years
  Responses of participants regarding concern of Multiple Sclerosis (MS) for next visit, priority and wellness goals, and how close they are completing the goal will be recorded.
Expanded Disability Status Scale (EDSS) Score | Baseline up to 3 years
Multiple Sclerosis Functional Composite (MSFC) Score | Baseline up to 3 years
Timed 25-Foot Walk Test | Baseline up to 3 years
9-Hole Peg Test (9HPT) Score | Baseline up to 3 years
Paced Auditory Serial Addition Test (PASAT) Score | Baseline up to 3 years
Symbol Digit Modalities Test (SDMT) | Baseline up to 3 years
Processing Speed Test (PST) | Baseline up to 3 years
Number of Participants with Magnetic resonance imaging (MRI) History | Baseline up to 3 years
Number of Participants with History of Fall | Baseline up to 3 years
Number of Participants with Adverse Events of Interest | Baseline up to 3 years
Number of Participants with Symptoms of Coronavirus (COVID) | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (9):
- United States (9):
  - Alabama Neurology Associates, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial healthcare, Owosso, Michigan
  - University of Nebraska medical Center, Omaha, Nebraska
  - The Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - The University of Texas of Austin, Austin, Texas
  - University of Texas Health, San Antonio, Texas

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200077_0021
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html